CLINICAL TRIAL: NCT01785550
Title: Ultrasonography in Amyotrophic Lateral Sclerosis as a Predictor of Disease Progression and Tool in Diagnosis: a Pilot Study
Brief Title: Neuromuscular Ultrasound in ALS
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00042025
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: ALS

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Group: No intervention to be performed.
- Ultrasound Group: All will receive nerve and muscle ultrasound.
  Interventions: Other: Ultrasound of nerve and muscle

INTERVENTIONS:
Other: Ultrasound of nerve and muscle — Ultrasound of 6 muscles and 2 nerves will be performed.
  Groups: Ultrasound Group

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is a progressive fatal neurodegenerative disease affecting motor neurons. Early diagnosis is essential for the success of clinical trials and objective biomarkers are needed for monitoring disease progression. Nerve and muscle ultrasound may provide this information.

This study will collect pilot data to evaluate the value of muscle and nerve ultrasound to identify and monitor disease progression in ALS.

ELIGIBILITY:
Inclusion Criteria:

* Subjects referred to the electromyography laboratory for ALS.

Exclusion Criteria:

* Patients with known comorbid myopathy or neuropathy will be excluded from the study.
* Patients unable to provide their own consent will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients referred to the electromyography laboratory for ALS.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Abnormalities at onset: Ultrasound vs. Electromyography | 1 year
  Ultrasound measures will be compared to electromyography measures at the patient's initial assessment. The number of abnormal muscles will be counted using each technique and analyzed to determine if one test is superior.

SECONDARY OUTCOMES:
Ultrasound Predicting Outcome at 1 year | 1.5 years
  The initial ultrasound measures and patient outcomes, as measured by standard validated scales, will be assessed at periodic intervals for one year. Analysis will be performed to determine if ultrasound measures can predict the clinical course.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States